CLINICAL TRIAL: NCT04269694
Title: Adjunctive Use of an Antibacterial Honey Dressing for Palatal Wound Healing After Harvesting a Free Gingival Graft: A Case-control Study
Brief Title: Adjunctive Use of an Antibacterial Honey Dressing for Palatal Wound Healing After Harvesting a Free Gingival Graft
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Riyadh Elm University (Other)
Responsible Party: Principal Investigator, Abdullah Alrashidi, Board periodontics resident, Riyadh Elm University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FPGRP/2019/438/36
Record Dates: First submitted 2020-02-10; First posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Healing Wound

STUDY DESIGN:
Intervention Model Description: In control group, no dressing material will be applied to donor site. While in test group, an antibacterial honey dressing material (Medihoney, http://www.medihoney.com) will be applied to donor site.
Masking Description: No masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Control (No Intervention): No dressing applied in the donor site after harvesting the graft
- Test (Experimental): An antibacterial honey dressing material (Medihoney, http://www.medihoney.com) will be applied to donor site.
  Interventions: Drug: Medihoney dressing; Device: Medihoney dressing

INTERVENTIONS:
Drug: Medihoney dressing — Medihoney is a mixture of two honeys derived from Australia and New Zealand containing glucose oxidase and Leptospermum compounds which contribute to its antibacterial activity.
  Other Names: K101793
  Arms: Test
Device: Medihoney dressing — Medihoney is a mixture of two honeys derived from Australia and New Zealand containing glucose oxidase and Leptospermum compounds which contribute to its antibacterial activity.
  Arms: Test

SUMMARY:
This case-control study will afford a more understanding of the clinically benefits that the antibacterial honey dressing material has in palatal wound healing and the subsequent effects in post-operative morbidity.

DETAILED DESCRIPTION:
Hard palate is considered the most common area to harvest a free gingival graft (FGG) for several periodontal plastic surgical procedures. Due to their autogenous nature, palatal grafts have excellent clinical results and are therefore superior to synthetic or allogenic grafts. An open wound at the donor site after harvesting the FGG takes two to four weeks to heal. Wound healing is a complex process containing various events. Firstly, the hemostatic phase which leads to sealing of the wound by a clot formed by platelets and other blood-derived cells in a network composed of fibrin, fibronectin, and vitronectin. Secondly, the inflammatory phase which advances a catabolic inflammatory process mediated by neutrophils and monocytes that leads to wound cleansing. Thirdly, the formation phase that originated by granulation tissue formation which is replaced by provisional connective tissue. Three major cell types are involved in this anabolic phase: (1) Endothelial cells and progenitors for the formation of capillaries. (2) Fibroblasts and myofibroblasts required for connective tissue formation and wound shrinkage. (3) Epithelial cells which contribute to re-epithelialization. Lastly, the remodeling phase which leaves a collagen-rich dense matrix containing a few cells that regenerates a stable tissue in the long term.

One of the possible complications after harvesting the FGG is the excessive post-operative morbidity which could be in the form of discomfort, pain and bleeding. These problems may affect patient quality of life and may disturb his/her daily activities such as eating, drinking or speaking. Therefore, it is of value to include patient-related outcomes in relation to quality of life measures after soft tissue grafts in clinical trials. Eltas et al. 2014 compared the effects of a periodontal dressing, the Essix retainer, the modified Essix retainer, and modified Hawley retainer on pain, chewing, speaking, and appearance. Using a periodontal dressing was associated with more pain and bleeding after one-week post-surgery; however, the speaking and appearance in the visual analog scale (VAS) scores were lower. In light of the above, retainers might be the most appropriate in terms of pain and bleeding, but less ideal for speaking and appearance comfort. In other studies, hyaluronic-acid gels as well as platelet-rich fibrin (PRF) were applied at the donor site after FGG harvesting. Both PRF and hyaluronic-acid may provide significant benefits for wound healing parameters and reduce pain. Keceli et al. 2015 evaluated the effectiveness of an herbal extract on early wound healing following FGG and found fewer incidences of primary and secondary bleeding as well as lower pain levels during the first postoperative week. In a human study Patel et al. 2012 demonstrated that ozonated oil was able to accelerate palatal wound epithelialization in a significant manner, compared with the control group.

Honey has been used for medicinal purposes since antiquity. Lee et al. 2011 noted that honey use for burn wounds has been documented in modern-day scientiﬁc journals since as early as 1933. As interest in honey for medical purposes grew, many FDA-approved products began emerging. With more interest came an increase in clinical studies examining honey for treatment of a variety of wounds, including randomized trials, case series, and cross-sectional studies from specialties ranging from dermatology and general surgery to ophthalmology.

Clinical parameters and procedures:

Patients will receive an initial periodontal examination and treatment, if necessary. Full-mouth plaque score and full-mouth bleeding score needed to be <20% to be eligible. Surgical procedures will be performed by the same periodontist. For all measurements the same periodontal probe (Hu-Friedy PCPUNC 15 mm, Hu-Friedy, Chicago, IL.) will be used. At the donor site, anesthesia will be achieved with palatal local inﬁltrations, with 1.8 mL lidocaine 2% 1:100,000 epinephrine. Once the graft is harvested, pressure will be applied to the palate until hemostasis is achieved. The length and width of the donor site will be measured and recorded. In control group, no dressing material will be applied to donor site. While in test group, an antibacterial honey dressing material (Medihoney, http://www.medihoney.com) will be applied to donor site. Medihoney is a mixture of two honeys derived from Australia and New Zealand containing glucose oxidase and Leptospermum compounds which contribute to its antibacterial activity. It is licensed for wound care in Australia, Europe and the USA. It works with the body's natural processes to bathe the wound bed promoting the removal of devitalized tissue. Its low pH (3.5-4.5) helps to lower the pH within the wound environment, which has been shown to have wound healing benefits.

All patients will receive the same analgesic (ibuprofen 600 mg) immediately after the surgery. All patients will receive the same postoperative instructions. Soft diet will be recommended for all patients. Chlorhexidine 0.12% mouth rinse will be prescribed to each patient for use twice daily. Ibuprofen 600 mg will also be prescribed for the patients to consume 1 tablet orally for every 8 hours. The participants will be asked to note the level of pain, and the level of discomfort (eating, speaking, etc.) from the donor site during the ﬁrst postoperative week using a 0 to 10 pain visual analog scale (VAS) score by graphic format. Discomfort was deﬁned as irritating sensation and diﬃculty in eating, speaking, etc. and pain as inability to function requiring analgesics. At the 1-week, 2-week and 4-week follow-up appointments, the length and width of the donor site will be measured and recorded.

ELIGIBILITY:
Inclusion Criteria:

* be 18 years and more
* systemically healthy
* non-smoker
* full-mouth plaque and bleeding scores <20%,

Exclusion Criteria:

* has history of mucogingival surgery on the palatal area
* pregnant women
* systemic antibiotics taken for at least six months
* has coagulation disorders (e.g. Hemophilia a/b, von Willebrand disease, liver disease, anticoagulative therapy)
* on corticosteroids, or with any systemic disease that precluded periodontal surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in length and width of the donor site | At the 1-week, 2-week and 4-week follow-up appointments
  Using periodontal probe (Hu-Friedy PCPUNC 15 mm, Hu-Friedy, Chicago, IL.)

SECONDARY OUTCOMES:
The level of pain and the level of discomfort | At the 1-week
  Using 0-10 visual analog scale (no pain on the left end (0) of the scale and the "worst pain" on the right end of the scale (10)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available

REFERENCES:
- [Background] Burkhardt R, Hammerle CH, Lang NP, Research Group on Oral Soft Tissue B, Wound H. (2015) Self-reported pain perception of patients after mucosal graft harvesting in the palatal area. J Clin Periodontol 42:281-287 Chaiken, N. (2010) Pressure ulceration and the use of Active Leptospermum honey for debridement and healing. Ostomy Wound Management 56(5), 12-14. Cortellini P, Pini Prato G. (2012) Coronally advanced flap and combination therapy for root coverage. Clinical strategies based on scientific evidence and clinical experience. Periodontol 2000 59:158-84. Eltas A, Eltas SD, Uslu MO, Ersöz M. (2014) Evaluation of patient discomfort at the palatal donor site following free gingival graft procedures: A randomized controlled clinical trial. J Periodontol Implant Dent. 6:47-53. Farnoush A. (1978) Techniques for the protection and coverage of the donor sites in free soft tissue grafts. J Periodontol. 49(8):403-5. Keceli HG, Aylikci BU, Koseoglu S, Dolgun A. (2015) Evaluation of palatal donor site haemostasis and wound healing after free gingival graft surgery. J Clin Periodontol. 42(6):582-9. Lee DS, Sinno S, Khachemoune A. (2012) Honey and wound healing: an overview. Am J Clin Dermatol. 12(3):181-90. Lorenzana ER, Allen EP. (2000) The single-incision palatal harvest technique: A strategy for esthetics and patient comfort. Int J Periodontics Restorative Dent. 20:297-305. Milne SD, Connolly P. (2014) The influence of different dressings on the pH of the wound environment. J Wound Care. 23(2):53-4, 56-7. Molan PC. (2006) The evidence supporting the use of honey as a wound dressing. Int J Low Extrem Wounds 5:40-54. Ozcan, M., Ucak, O., Alkaya, B., Keceli, S., Seydaoglu, G., & Haytac, M. C. (2017) Effects of Platelet-Rich Fibrin on Palatal Wound Healing After Free Gingival Graft Harvesting: A Comparative Randomized Controlled Clinical Trial. International Journal of Periodontics & Restorative Dentistry, 37(5). Patel PV, Kumar S, Vidya GD, Patel A, Holmes JC, Kumar V. (2012) Cytological assessment of healing palatal donor site wounds and grafted gingival wounds after application of ozonated oil: an eighteen-month randomized controlled clinical trial. Acta Cytol. 56(3):277-84. Yıldırım S, Özener HÖ, Doğan B, Kuru B. (2017) Effect of topically-applied hyaluronic-acid on pain and palatal epithelial wound healing: An examiner-blind, randomized, controlled clinical trial. J Periodontol. 88:1-14. Zucchelli G, Mele M, Stefanini M, Mazzotti C, Marzadori M, Montebugnoli L, et al. (2010) Patient morbidity and root coverage outcome after subepithelial connective tissue and de-epithelialized grafts: A comparative randomized-controlled clinical trial. J Clin Periodontol 37:728-38.